CLINICAL TRIAL: NCT00230282
Title: A Multi-Center Phase 2 Efficacy and Pharmacokinetic Study Evaluating Fludarabine, Cyclophosphamide, and Subcutaneous Campath (FCCam, Alemtuzumab) for Previously Untreated B-Cell Chronic Lymphocytic Leukemia
Brief Title: Phase 2 Fludarabine, Cytoxan and FCCAM <Alemtuzumab> in Untreated B-Cell Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Steven E. Coutre (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor-Investigator, Steven E. Coutre, Associate Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-13053; 31185 (Other: Berlex Oncology ID); 80071 (Other: Stanford University Alternate IRB Approval Number); HEMCLL0001 (Other: OnCore)
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-09

CONDITIONS: Leukemia; B-cell Leukemia; Chronic Leukemia; Chronic Lymphocytic Leukemia (CLL)
MeSH Terms: conditions — Leukemia; Leukemia, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Alemtuzumab; fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fludarabine, cytoxan, then alemtuzumab (Experimental): Fludarabine and cyclophosphamide days 1 to 3 for six 28-day cycles. Minimal residual disease positive responders continued on-treatment to receive alemtuzumab 30 mg weekly. MRD negative responders were observed.
  Interventions: Drug: Alemtuzumab; Drug: Fludarabine; Drug: Cytoxan

INTERVENTIONS:
Drug: Alemtuzumab — 3 to 30 mg, IV
  Other Names: Campath; MabCampath; Campath-1H; Lemtrada; FCCam
Drug: Fludarabine — [(2R,3R,4S,5R)-5-(6-amino-2-fluoro-purin-9-yl)- 3,4-dihydroxy-oxolan-2-yl]methoxyphosphonic acid
  Other Names: Fludara
Drug: Cytoxan — (RS)-N,N-bis(2-chloroethyl)-1,3,2-oxazaphosphinan-2-amine 2-oxide
  Other Names: Cyclophosphamide; cytophosphane; Endoxan; Neosar; Procytox; Revimmune

SUMMARY:
The primary objective of this study was to evaluate the safety and efficacy of the combination of fludarabine and cyclophosphamide in previously untreated CLL patients. Participants will receive fludarabine and cyclophosphamide on days 1, 2, and 3 of six 28-day cycles.

DETAILED DESCRIPTION:
This single-arm study evaluated the safety and efficacy of the combination of fludarabine 25 mg/m2/d IV and cyclophosphamide 250 mg/m2/d SC in previously untreated CLL patients. Participants received fludarabine and cyclophosphamide on days 1, 2, and 3 of six 28-day cycles, followed by a no-treatment rest period (observation) for 3 to 12 weeks.

Responders entered a no-treatment rest period (observation) for 3 to 8 weeks, then depending on status, continued on follow-up or on-study to receive Campath stating at 3 mg/day with the dose adjusted to the maximum tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

* ≥ age 18
* Karnofsky performance status 60% or above
* Confirmed immunohistological diagnosis of Chronic Lymphocytic Leukemia (CLL)
* Rai Stage I to IV as follows:

  * Advanced stage disease (Rai Stage III or IV, or modified Rai High Risk)
  * OR
  * Patients with Rai Stage I - II or (Modified Rai Intermediate-Risk) disease must have an indication for therapy based on 1996 NCI revised criteria for active disease as follows:

    * Any one of the following disease-related symptoms:

      1. Weight loss ≥ 10% body weight within the previous 6 months
      2. Extreme fatigue
      3. Fever greater than 100.5° F for ≥ 2 weeks without evidence of infection
      4. Night sweats without evidence of infection
    * Evidence of progressive marrow failure based on the development of worsening of anemia or thrombocytopenia
    * Autoimmune anemia and/or thrombocytopenia poorly responsive to corticosteroid therapy
    * Massive (> 6 cm below the left costal margin) or progressive splenomegaly
    * Bulky (>10 cm in cluster) or progressive lymphadenopathy
    * Progressive lymphocytosis > 50% increase over 2 months, or anticipated doubling time < 6 months
* Patients with immunoglobulin VH gene in unmutated nucleotide sequence configuration, as defined by ≥ 98% homology with the nearest germline counterpart
* Serum creatinine ≤ 2x the upper limit of normal
* Total serum bilirubin ≤ 2x the upper limit of normal.
* AST ≤ 2x the upper limit of normal.
* ALT ≤ 2x the upper limit of normal.
* Signed written informed consent

Exclusion Criteria:

* Prior pharmacological treatment for CLL
* Past history of anaphylaxis following exposure to monoclonal antibodies
* Active secondary malignancy or a history of malignant disease (other than CLL or non-melanoma skin cancer) within the preceding 5 years
* Any medical condition requiring systemic corticosteroids
* Active systemic infection
* Major systemic or other illness (including Coombs positivity and active hemolysis) that would, in the opinion of the investigator, interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of study results
* HIV positive by serologic testing
* Pregnant or nursing female
* Unwilling/unable to practice an acceptable form of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-07; Primary Completion 2010-12 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Edward Coutre, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fludarabine and Cyclophosphamide, Followed by Alemtuzumab: Fludarabine 25 mg/m2/d IV and cyclophosphamide 250 mg/m2/d SC on days 1 to 3 for each of six 28-day cycles, when the assessment for Primary Completion occurred. Responders entered a no-treatment rest period (observation) for 3 to 8 weeks, then depending on status, continued on follow-up or on-study to receive alemtuzumab IV starting at 3 mg/day with the dose adjusted to the maximum tolerated dose (up to 30 mg).
Period: Fludarabine + Cyclophosphamide
Arm/Group | Fludarabine and Cyclophosphamide, Followed by Alemtuzumab
Started | 25
Completed | 17
Not Completed | 8
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 1
Not completed — Change in diagnosis | 1
Not completed — Richters transformation (progression) | 2
Period: Maintanence Therapy With Alemtuzumab
Arm/Group | Fludarabine and Cyclophosphamide, Followed by Alemtuzumab
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fludarabine and Cyclophosphamide, Followed by Alemtuzumab
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Maintaining Partial Response (PR) or Complete Response (CR)
Description: Response criteria as per the NCI-WG Revised Guidelines for B-CLL
  Complete remission:
  No lymphadenopathy by physical exam No hepatomegaly or splenomegaly Absence of constitutional symptoms Polymorphonuclear leukocytes > 1,500/uL, Platelets > 100,000/uL, Hemoglobin > 11.0 g/dL Bone marrow aspirate and biopsy normocellular with < 30% lymphocytes Absent lymphoid nodules
  Partial remission:
  * 50% decrease in peripheral blood lymphocyte count from the pretreatment baseline value
  * 50% reduction in lymphadenopathy and/or ≥ 50% reduction in the size of the liver and/or spleen AND one or more of the following Polymorphonuclear leukocytes > 1,500/uL or 50% improvement over baseline Platelets > 100,000/uL or 50% improvement over baseline Hemoglobin > 11.0 g/dL or 50% improvement over baseline
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Fludarabine and Cyclophosphamide, Followed by Alemtuzumab
Number analyzed (Participants) | 25
participants | 17

2. Secondary Outcome: Duration of Response
Time Frame: 105 months
Measure: Median (Full Range); unit: months
Arm/Group | Fludarabine and Cyclophosphamide, Followed by Alemtuzumab
Number analyzed (Participants) | 17
months | 38 [12 to 105]

ADVERSE EVENTS:
Arm/Group | Fludarabine, Cytoxan, Then Alemtuzumab
Serious Adverse Events (participants affected / at risk) | 5/25
Other Adverse Events (participants affected / at risk) | 2/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fludarabine, Cytoxan, Then Alemtuzumab (N=25)
febrile neutropenia (Blood and lymphatic system disorders) | 1 — G3; hospitalization after 4th cycle. Resolved with empiric antibiotics.
anemia (Blood and lymphatic system disorders) | 1 — G3; required transfusion. Pre-existing AIHA
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 — G3 Required brief course of oxygen therapy
lung infection (Infections and infestations) | 1 — G3 Hospitalized. Received IV antibiotics with resolution.
hemolysis (Blood and lymphatic system disorders) | 1 — G3. Pre-existing AIHA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fludarabine, Cytoxan, Then Alemtuzumab (N=25)
anemia (Blood and lymphatic system disorders) | 1 — G3
mucositis (Gastrointestinal disorders) | 1 — G3 Oral mucositis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No